CLINICAL TRIAL: NCT06001515
Title: Effect of Face Scanning on Accuracy of Dental Implant Placement in Fixed Implant Supported Maxillary Prostheses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Abdelmoez, assistant lecturer of oral and maxillofacial prosthodontics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-RecID012328
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Computer-Assisted Surgery
Keywords: guided implant placement- face scanning - edentulous maxilla

STUDY DESIGN:
Intervention Model Description: one experimental group and one active comparator group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual scan protocol (Active Comparator): Two CBCT scans will be made.One while the patient wearing the radiographic stent and another CBCT for the radiographic stent alone.
  Interventions: Device: Dual scan protocol
- Dual scan protocol +3D facial scan record (Experimental): 3D face scan record will be made plus Two CBCT scans. One while the patient wearing the radiographic stent and another CBCT for the radiographic stent alone.
  Interventions: Device: triple scan protocol

INTERVENTIONS:
Device: Dual scan protocol — one CBCT scan for the patient while wearing the scan appliance and another scan for the appliance alone
  Arms: Dual scan protocol
Device: triple scan protocol — 3D facial Scanning for the patients while wearing their dentures in addition to the dual scan protocol
  Arms: Dual scan protocol +3D facial scan record

SUMMARY:
The study will compare the accuracy of surgical guides fabricated by two different scanning protocols; facially driven scanning versus dual scanning protocol regarding the deviation of implant placement.

DETAILED DESCRIPTION:
Twelve completely edentulous patients will be selected for full arch maxillary guided implants placement with immediately loaded restoration. The patients will make a complete oral and radiographic examination before inclusion in this study. All patients will receive maxillary and mandibular complete dentures that will be made in a conventional way. The patients will be randomly divided into two equal groups; group (I) and group (II). In both groups two CBCT scans will be made. A CBCT scan will be made for each patient while wearing the radiographic stent and another CBCT scan will be made for the radiographic stent alone. However, for patients in group II a face scan will be added to previous scans. For each patient in group I, the DICOM files will be exported to Blue Sky implant designing software (Langenhagener, Mdi Europa GmbH), fusion of the scan prosthesis via the markers is accomplished and the ideal surgical site and optimal implant dimensions will be selected. All the surgical guides will be planned to be totally limiting in this study. The immediate provisional restoration will be planned on the software according to the previously planned implants sites. The surgical guide will be 3D printed. The approved tooth arrangement will be subsequently sent as an STL file to a milling machine. For each patient in group II, the DICOM files and the STL files obtained from the face scans will be exported to Blue Sky implant designing software (Langenhagener, Mdi Europa GmbH). The facial scan will be used to define the interpupillary and midsagittal planes and to examine the tooth form and buccal corridor width with regard to the patient's smile line. Both files data will be superimposed and the planning for the implants sites, surgical guide and immediate restoration will be done as in group I. After implant insertion, CBCT scan will be made for each patient while wearing the scan appliance. Superimposition of CBCT scans pre and post implant insertion and restoration will be made. Deviations between planned and placed implant will be measured in the lateral apical, lateral coronal and angular aspects. Also, the patient satisfaction will be measured on a likert scale.

ELIGIBILITY:
Inclusion Criteria:

- The inclusion criteria will be completely edentulous patients, non-smokers, 50-70 years in age, have Good oral hygiene and motivation.

Exclusion Criteria:

* The excluded patients will include patients with major systemic diseases that may affect osseointegration as uncontrolled diabetes mellitus, the need for extensive bone grafting in planned implant site, pregnancy, patients under bisphosphonate treatment, and limited mouth-opening for executing the guided implant surgery.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
( Assessment of linear deviation | 1day
  Accurate details recorded by superimposition of CBCTs using the blue sky software program by measuring the lateral coronal deviation in millimeters.
( Assessment of linear deviation | 1day
  Accurate details recorded by superimposition of CBCTs using the blue sky software program by measuring the lateral apical deviation in millimeter.
( Assessment of angular deviation | 1day
  Accurate details recorded by superimposition of CBCTs using the blue sky software program by measuring the angular deviation in degrees.

SECONDARY OUTCOMES:
patient satisfaction | 1 day
  Accurate details recorded by using a 5 points likert scale for measuring the patient satisfaction by filling specific questionnaire: Oral Health Impact Profile 14 questions ( OHIP-14) and taking the answer of each question on a 5 point likert scale with 0 for the worst score and 5 for the best one

CONTACTS AND LOCATIONS:
Overall Officials: Noha H Nawar, BDS MSc MD, Study Director — Ain Shams University
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Egypt